CLINICAL TRIAL: NCT00048139
Title: An Open-label Study of the Effect of Intermittent Xeloda in Combination With Irinotecan on Treatment Response in Patients With Advanced and/or Metastatic Colorectal Cancer
Brief Title: A Study of Xeloda (Capecitabine) in Patients With Advanced and/or Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO16461
Record Dates: First submitted 2002-10-24; First posted 2002-10-25 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Capecitabine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Irinotecan; Drug: capecitabine [Xeloda]

INTERVENTIONS:
Drug: Irinotecan — 250mg/m2 iv on day 1 of each 3 week cycle
Drug: capecitabine [Xeloda] — 1000mg/m2 po bid on days 1-15 of each 3 week cycle

SUMMARY:
This study will assess the efficacy and safety of intermittent oral Xeloda administration in combination with irinotecan as a first-line treatment in patients with advanced and/or metastatic colorectal cancer. The anticipated time on study treatment is 3-12 months and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* locally advanced and/or metastatic colorectal cancer;
* >=1 target lesion.

Exclusion Criteria:

* previous treatment with Xeloda or irinotecan;
* previous systemic therapy for metastatic disease;
* progressive disease during previous adjuvant therapy or within 6 months of completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2001-10; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Tumor measurement (RECIST criteria) | Event driven

SECONDARY OUTCOMES:
Efficacy: Time to progression, time to response, duration of response, time to treatment failure, survival. | Event driven

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- United States (10):
  - Phoenix, Arizona
  - Fountain Valley, California
  - La Jolla, California
  - Santa Rosa, California
  - Denver, Colorado
  - Hutchinson, Kansas
  - Las Vegas, Nevada
  - Albuquerque, New Mexico
  - Buffalo, New York
  - Houston, Texas